CLINICAL TRIAL: NCT02179775
Title: Comparison of Effectiveness of "Sekanjabin e Safarjali" (Quince Oxymel), Propranolol and Placebo in the Prevention of Migraine Attacks in Patients With Simultaneous Upper Gastrointestinal Dysfunction
Brief Title: Effect of "Sekanjabin e Safarjali" (Quince Oxymel) in the Prevention of Migraine Attacks
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mohammad Hashem Hashempur, MD, PhD of Iranian traditional medicine, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 90-01-64-3456
Record Dates: First submitted 2014-06-27; First posted 2014-07-02 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-07

CONDITIONS: Migraine Headache; Gastric Diseases
MeSH Terms: conditions — Migraine Disorders; Stomach Diseases | interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- propranolol (Active Comparator)
  Interventions: Drug: propranolol
- Quince's oxymel (Active Comparator)
  Interventions: Drug: Quince's oxymel
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: propranolol
  Arms: propranolol
Drug: Quince's oxymel
  Arms: Quince's oxymel
Drug: placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to determine whether Quince Oxymel is effective in the prevention of Migraine attacks in patients with simultaneous upper gastrointestinal dysfunction.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, triple blinded clinical study to evaluate the effects of oral use of "Sekanjebin e Safarjali" (Quince Oxymel) in the Prevention of Migraine attacks in patients with simultaneous upper gastrointestinal dysfunction.45 patients with Migraine headache aged between 15-70, after taking signed informed consent, according to the International headache society criteria for headache [2] are included in this trial. 45 cases with Migraine headache with simultaneous upper gastrointestinal dysfunction will allocate to three arms by using simple randomization. Quince Oxymel, propranolol and placebo will be given as encoded, innominate bottles with the same shape and color. Quince oxymel and placebo will be prescribed as 10 cc, three times a day for 4 weeks. Frequency, duration and intensity of Migraine Attacks at the beginning time and during 4 weeks of trial, will be evaluated, as the primary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* minimum age of 18 years old
* giving a written informed consent
* having at least 2 migraine attacks per month

Exclusion Criteria:

* patients older than 70 years old
* patients with Diabetes mellitus
* patients with chronic obstructive pulmonary disease and asthma
* pregnancy
* severe depression
* patients affected by sexual disorders
* bradyarrhythmic patients
* positive history of hypersensitivity reactions to quince, ginger, propranolol or naproxen

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2014-07; Primary Completion 2014-09 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
frequency of headache attacks | 4 weeks
duration of headache attacks | 4 weeks
Pain Scores as assessed by the Visual Analog Scale | 4 weeks

SECONDARY OUTCOMES:
self-reported improvement of upper gastrointestinal symptoms (by percent) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Abdolhamid Shariat, MD, Assistant Professor, Principal Investigator — Shiraz University of Medical Sciences
Locations (1):
- Shiraz University of Medical Sciences, Shiraz, Fars, Iran